CLINICAL TRIAL: NCT07267455
Title: Efficacy Analysis of Personalized-Target Transcranial Magnetic Stimulation (TMS) in the Treatment of Chronic Tinnitus: A Single-Center, Single-Blind Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2025-648-02
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Chronic Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized-Target TMS Group (Experimental): Participants receive continuous theta burst stimulation (cTBS) targeting the individualized auditory cortex region showing the strongest functional connectivity with the left parahippocampal gyrus, as identified by resting-state fMRI. Each participant receives 600 pulses per session, 3 sessions per day (total 1,800 pulses daily) for 5 consecutive days.
  Interventions: Device: continuous theta burst stimulation
- conventional auditory cortex site (Active Comparator): Participants receive continuous theta burst stimulation (cTBS) targeting the left auditory cortex at EEG 10-20 system site CP5, as used in prior tinnitus studies. Stimulation parameters are identical to the experimental group (600 pulses per session, 3 sessions per day, for 5 consecutive days).
  Interventions: Device: continuous theta burst stimulation

INTERVENTIONS:
Device: continuous theta burst stimulation — This study evaluates personalized-target and conventional-target transcranial magnetic stimulation (TMS) for the treatment of chronic subjective tinnitus. Participants will receive continuous theta burst stimulation (cTBS) applied to the left auditory cortex. For the personalized-target arm, stimulation sites are individualized based on resting-state fMRI, targeting the region of strongest functional connectivity with the parahippocampal gyrus. For the conventional-target arm, stimulation is delivered at the CP5 site. Each session consists of 600 pulses, delivered in three sessions per day (1,800 pulses daily) for five consecutive days.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of personalized-target transcranial magnetic stimulation (TMS) in the treatment of chronic subjective tinnitus. The study aims to determine whether stimulation at individualized auditory cortex targets, identified by resting-state functional MRI, provides greater therapeutic benefit compared with conventional TMS targets.

A total of 116 patients with chronic tinnitus will be recruited and randomly assigned to receive either personalized-target TMS or traditional-target TMS for five consecutive days.

The main questions this study aims to answer are:

Does personalized-target TMS improve tinnitus-related symptoms more effectively than traditional-target TMS?

Is personalized-target TMS a safe and tolerable intervention for patients with chronic tinnitus?

Researchers will compare the changes in tinnitus-related clinical rating scales between the two groups, including the Tinnitus Handicap Inventory (THI), Visual Analog Scale (VAS), Beck Anxiety Inventory (BAI), Beck Depression Inventory (BDI), and Pittsburgh Sleep Quality Index (PSQI).

Participants will:

Receive continuous theta burst stimulation (cTBS) targeting the left auditory cortex region showing the strongest functional connectivity with the parahippocampal gyrus, identified through resting-state fMRI.

Undergo three cTBS sessions per day (600 pulses per session, 1,800 pulses total daily) for five days.

Complete follow-up assessments at 1 month and 3 months after treatment to evaluate the durability of clinical effects.

This study will also assess treatment adherence, safety outcomes, and potential predictors of therapeutic response to personalized-target TMS.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with tinnitus as the main complaint: Patients perceive subjective sounds in the ears or deep within the skull in the absence of internal or external acoustic stimulation.

  2.Patients with chronic tinnitus who meet the conditions including tinnitus duration of more than 6 months, THI (tinnitus handicap inventory) score ≥ 38, and no response to conventional drug treatment.

  3.Outpatients of Sun Yat-sen University Sun Yat-sen Memorial Hospital who can receive continuous 5-day cTBS treatment.

  4.Tinnitus frequency ranges from 125 Hz to 8000 Hz. 5.Aged 18-70 years.

Exclusion Criteria:

* 1.Patients with tinnitus associated with the following conditions: conductive hearing loss, a history of middle ear surgery, pulsatile tinnitus caused by vascular malformations, or Meniere's disease.

  2.A history of any of the following: head trauma, central nervous system diseases, psychiatric disorders, or substance abuse.

  3.Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 116 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
the effective rate of chronic tinnitus relief in the two groups of patients before treatment and 5 days after treatment | From enrollment to the end of treatment at 5 days
  It is defined as follows:
  Effective rate = [(Number of patients in each group who completed the 5-day treatment and had a Tinnitus Handicap Inventory (THI) score decrease of ≥ 7 points from the baseline) / (Total number of patients in each group who completed the 5-day treatment)] × 100%. The assessment time points for this outcome are before treatment (baseline) and 5 days after treatment.

SECONDARY OUTCOMES:
Tinnitus Loudness | Baseline, post-treatment (day 5), 1-month follow-up, 3-month follow-up
  Change in tinnitus loudness, assessed using the Visual Analog Scale (VAS), which ranges from 0 (no tinnitus) to 10 (worst tinnitus imaginable).
Anxiety Symptoms | Baseline, post-treatment (day 5), 1-month follow-up, 3-month follow-up
  Change in anxiety symptoms, assessed using the Beck Anxiety Inventory (BAI), a self-reported questionnaire measuring severity of anxiety.
Depressive Symptoms | Baseline, post-treatment (day 5), 1-month follow-up, 3-month follow-up
  Change in depressive symptoms, assessed using the Beck Depression Inventory (BDI), a self-reported scale evaluating severity of depression.
Sleep Quality | Baseline, post-treatment (day 5), 1-month follow-up, 3-month follow-up
  Change in sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI), which evaluates sleep quality and disturbances over a 1-month period.
Long-term Efficacy of Tinnitus Relief | 1-month follow-up, 3-month follow-up
  Effective rate = [(Number of patients in each group who completed the 5-day treatment and had a Tinnitus Handicap Inventory (THI) score decrease of ≥ 7 points from the baseline) / (Total number of patients in each group who completed the 5-day treatment)] × 100%. The assessment time points for this outcome are before treatment (baseline) and 1 month, 3 month after treatment.
EEG Changes | Baseline (pre-treatment), post-treatment (day 5), 1-month follow-up, 3-month follow-up
  Changes in electroencephalography (EEG) measures associated with tinnitus and cortical activity, assessed before treatment, after 5 days of intervention, and at 1-month and 3-month follow-ups.
MRI Changes | Baseline (pre-treatment), 1-month follow-up
  Changes in brain structure and functional connectivity assessed using magnetic resonance imaging (MRI), including the auditory cortex and related networks. MRI is performed at baseline (pre-treatment) and at 1-month follow-up to evaluate early post-treatment neural changes.

CONTACTS AND LOCATIONS:
Overall Officials: Yuexin Cai, Doctor, Study Chair — Yuexin Cai, Doctor
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to privacy concerns and ethical restrictions related to patient confidentiality.